CLINICAL TRIAL: NCT05321979
Title: Open-label, Single Group, Multi-center, Repeat-dose Long-term Extension Study to Evaluate the Long-term Safety and Efficacy of MBA-P01 in Subjects With Moderate to Severe Glabellar Lines
Brief Title: Long-term Extension Study to Evaluate MBA-P01 in Subjects With Moderate to Severe Glabellar Lines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medytox Korea (Industry)
Responsible Party: Sponsor
Organization: Medy-Tox (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT14-KR21GBL1202
Record Dates: First submitted 2022-03-23; First posted 2022-04-11 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Glabellar Frown Lines

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MBA-P01 (Experimental): MBA-P01 will be injected into GL:
  Interventions: Drug: MBA-P01

INTERVENTIONS:
Drug: MBA-P01 — MBA-P01 will be injected into the Glabellar line.

SUMMARY:
This study is intended to evaluate long-term safety and efficacy of MBA-P01 in treatment of glabellar lines.

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed the phase III trial (MT14-KR20GBL309)
* Patients who were capable of understanding and complying with the protocol and have signed the informed consent form voluntarily

Exclusion Criteria:

* Patients who have received other procedures which may affect glabellar lines within 6 months (except of MBA-P01 or BOTOX® treated in phase III trial, MT14-KR20GBL309)
* Female patients who are pregnant or lactating. Female patients of childbearing age who have a plan to get pregnant during the study period.
* Patient who do not use available contraceptive methods (Women of childbearing age should have negative urine pregnancy test results at baseline visit (0 week) prior to the first injection.)
* Patients who are participating in other clinical trials or have participated in other clinical trials 30 days before screening
* Patients who are not eligible for this study based on the judgment of an investigator

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Incidence rate of treatment-emergent adverse events (TEAEs), adverse drug reactions (ADRs), serious adverse events (SAEs) and adverse event of special interest (AESI), when MBA-P01 is administered in repeated treatments. | Through study completion, an average of 1 year
Incidence rate of TEAE, ADR, SAE and AESI of each cycle | Through each cycle, an average of 3 months
The change of laboratory test and vital sign | Through study completion, an average of 1 year
The result of anti-drug-andibodies (ADA) and neutralizing antibodies | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
Investigator-rated improvement rate of glabellar lines (GL) at maximum frown at week 4, week 8 and 12 of each cycle | at week 4, week 8 and 12 of each cycle
  Proportion of paricipants achieving at least a 2-grade improvement from reatreatment day and a grade 0 (none) or 1 (mild) in GL severity* as assessed by investigator
  *GL severity: 0=none, 1=mild, 2=moderate, 3=severe
Investigator-rated improvement rate of GL at rest at week 4, week 8 and 12 of each cycle | at week 4, week 8 and 12 of each cycle
  Proportion of participants who were grade 2 (moderate) on retreatment day and achieving grade 0 (none) or 1 (mild) at week 4, week 8 and 12 in GL severity* as assessed by investigator
  *GL severity: 0=none, 1=mild, 2=moderate, 3=severe
Participant-rated improvement rate of GL at frown at week 4, week 8 and 12 of each cycle | at week 4, week 8 and 12 of each cycle
  Proportion of participants achieving at least a 2-grade improvement from reatreatment day and a grade 0 (none) or 1 (mild) in GL severity* as assessed by participant
  *GL severity: 0=none, 1=mild, 2=moderate, 3=severe
Participant-rated improvement rate of GL at rest at week 4, week 8 and 12 of each cycle | at week 4, week 8 and 12 of each cycle
  Proportion of participants who were grade 2 (moderate) on retreatment day and achieving grade 0 (none) or 1 (mild) at week 4, week 8 and 12 in GL severity* as assessed by participant
  *GL severity: 0=none, 1=mild, 2=moderate, 3=severe
Participant-rated satisfaction rate of GL at rest at week 4, week 8 and 12 of each cycle | at week 4, week 8 and 12 of each cycle
  Participant evaluate the level of safisfaction by 7-grade score
Time to retreatment | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-Ang Univ. Hospital, Seoul, Dongjak-gu, South Korea

REFERENCES:
- [Derived] Han HS, Kim WS, Lee YW, Won CH, Lee W, Choi SY, Kim BJ. Long-term safety and efficacy of MBA-P01 for the treatment of glabellar lines: results from a multicenter, repeated-dose, open-label extension study. J Dermatolog Treat. 2024 Dec;35(1):2418919. doi: 10.1080/09546634.2024.2418919. Epub 2024 Oct 27. PMID 39462517